CLINICAL TRIAL: NCT03556007
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Ascending Multiple-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous NKTR-358 in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of NKTR-358 (LY3471851) in Participants With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17238; J1P-MC-KFAB (Other: Eli Lilly and Company); 17-358-02 (Other: Nektar Therapeutics)
Record Dates: First submitted 2018-05-07; First posted 2018-06-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Systemic Lupus Erythematosus
Keywords: T regulatory cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - 3 μg/kg LY3471851 (Experimental): Participants received 3 microgram per kilogram (μg/kg) of LY3471851 or placebo on days 1, 15 and 29 by subcutaneous (SC) injection.
  Interventions: Drug: LY3471851; Drug: Placebo
- Cohort 1 - 6 μg/kg LY3471851 (Experimental): Participants received 6 μg/kg of LY3471851 or placebo on days 1, 15 and 29 by SC injection.
  Interventions: Drug: LY3471851; Drug: Placebo
- Cohort 1 - 12 μg/kg LY3471851 (Experimental): Participants received 12 μg/kg of LY3471851 or placebo on days 1, 15 and 29 by SC injection.
  Interventions: Drug: LY3471851; Drug: Placebo
- Cohort 1 - 24 μg/kg LY3471851 (Experimental): Participants received 24 μg/kg of LY3471851 or placebo on days 1, 15 and 29 by SC injection.
  Interventions: Drug: LY3471851; Drug: Placebo

INTERVENTIONS:
Drug: LY3471851 — LY3471851 drug product is a sterile liquid for subcutaneous injection that will be diluted with sterile 0.9% sodium chloride solution for injection (USP) prior to administration.
  Other Names: NKTR-358
Drug: Placebo — The placebo dosing solution is 0.9% sodium chloride for injection (USP).

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of a study drug known as LY3471851 in participants with SLE. The study will last about 79 days for each participant.

DETAILED DESCRIPTION:
LY3471851 is a potential first-in-class therapeutic that may address an underlying immune system imbalance in people with many autoimmune conditions. It targets the interleukin (IL-2) receptor complex in the body in order to stimulate proliferation of inhibitory immune cells known as regulatory T cells. By activating these cells, LY3471851 may act to bring the immune system back into balance.

This study will evaluate the safety, tolerability, pharmacokinetics (PK), and immunologic effects of multiple doses of LY3471851 in participants with minimal to moderate SLE. The effects on SLE disease activity will also be evaluated. SLE participants will be randomized to receive multiple subcutaneous (SC) doses of LY3471851 or receive placebo. After receiving the last dose of LY3471851 or placebo, participants will be followed for an additional 50 days to evaluate safety, PK, pharmacodynamics (PD), and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent and comply with study procedures and requirements.
* Body mass index (BMI) between 18.0 and 32.0 kilograms per square meter (kg/m²).
* Systolic blood pressure between 90 to 140 millimeters of mercury (mm Hg), diastolic blood pressure between 50 to 90 mm Hg, and resting heart rate between 40 to 100 beats per minute.
* Diagnosis of adult SLE according to the 1997 ACR classification criteria for at least 6 months prior to signing the informed consent form (ICF).
* Minimal to moderate SLE disease activity (active SLE clinical disease is not required for enrollment into the study and participants with severe SLE clinical disease activity, based on the evaluation of the investigator, should be excluded).
* If a participant is taking oral prednisone (or prednisone equivalent) for their SLE, the dose must be less than or equal to (≤) 10 milligrams per day (mg/day) for a minimum of 8 weeks prior to screening. In addition, the dose of oral prednisone or prednisone equivalent the participant is taking must be stable for a minimum of 2 weeks prior to screening.
* If a participant is taking any of the medications below for their SLE, the medication must have been administered for a minimum of 12 weeks prior to signing the ICF, and at a stable dose for a minimum of 8 weeks prior to signing the ICF:

  * Azathioprine ≤ 200 mg/day
  * Antimalarial (e.g., chloroquine, hydroxychloroquine, quinacrine)
  * Mycophenolate mofetil ≤ 2 grams per day (g/day) or mycophenolic acid ≤ 1.44 g/day
  * Oral, SC, or intramuscular methotrexate ≤ 15 milligrams per week (mg/week).
* Willing and able to participate in the study for a duration of up to 4 months.
* Willing and able to abstain from participating in another clinical study for a duration of up to 4 months.
* Female participants will be non-pregnant, non-lactating, and either postmenopausal for at least 2 years, or surgically sterile for at least 3 months, or will agree to use double barrier contraception from period prior to study enrollment until 5 months following the last dose received; women of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) test at screening and randomization prior to administration of investigational product.
* Male participants with female partners of childbearing potential must agree to use double barrier contraception during the study (until 5 months following the last dose received). Sperm donation is also restricted during the time-frame that males must be using double barrier contraception. This criterion may be waived for male participants who have had a vasectomy greater than (>) 6 months prior to enrollment.

Exclusion Criteria:

Medical Conditions:

* Current active bacterial, viral, or fungal infection.
* Evidence of significant hematologic dysfunction.
* Evidence of significant liver or kidney dysfunction.
* History of, or current diagnosis of, a clinically significant non SLE-related vasculitis syndrome.
* Active severe or unstable neuropsychiatric SLE.
* Active severe SLE-driven renal disease or history of severe active lupus nephritis with persisting proteinuria levels greater than 0.5 grams/24 hours.
* Diagnosis (within 1 year of signing the ICF) of mixed connective tissue disease or any history of overlap syndromes of SLE.
* History of, or current, inflammatory joint or skin disease other than SLE.
* History of any non-SLE disease that has required treatment with oral or parenteral corticosteroids for more than 2 weeks within the last 24 weeks prior to signing the ICF.
* Active tuberculosis (TB) on the basis of positive medical history or chest radiograph (OR) evidence of latent TB or by positive (or persistently indeterminate) Quantiferon-TB Gold or T-Spot test.
* Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection.
* Confirmed positive serology for hepatitis B, hepatitis C (Viral Hepatitis C Antibody Screen [anti-HCV]), or a positive result for human immunodeficiency virus (HIV) antibody screen.
* Any severe herpes infection at any time prior to screening per judgement of the investigator.
* History of opportunistic infection requiring hospitalization or intravenous antimicrobial treatment within 3 years prior to randomization.
* History of major surgery within 12 weeks of screening or will require major surgery during the study.
* Clinically significant electrocardiographic abnormalities.
* History of any significant cardiovascular disease (e.g., myocardial infarction, congestive heart failure, uncontrolled hypertension, cerebrovascular accident), thrombotic episode, or any severe non-SLE medical illness within the previous 1 year.
* History of cancer, apart from:

  * Squamous or basal cell carcinoma of the skin that has been successfully treated.
  * Cervical cancer in situ that has been successfully treated.

Medications:

* Receipt of any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives prior to signing of the ICF, whichever is greater.
* Receipt of belimumab in 6 months prior to screening.
* History of treatment with rituximab or ocrelizumab (or other B cell depleting agent) within 6 months prior to screening. For participants who received their last treatment with rituximab or ocrelizumab more than 6 months earlier, evidence of significant and persisting low B cell levels in blood.
* History of cytotoxic medications (e.g., cyclophosphamide) within preceding 12 months.
* Receipt of any intra-articular, intramuscular, or intravenous (IV) glucocorticoids within 6 weeks prior to screening.
* Receipt of blood products within 6 months prior to screening.

General:

* Receipt of blood products within 6 months prior to screening and donation of blood or plasma to a blood bank or for a clinical study (except for screening of this study) within 28 days prior to screening.
* Participants who have a history of organ or bone marrow transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of LY3471851 - Number of Participants Experiencing Adverse Events | Informed consent until last study visit (approximately 79 days after first dose of study drug)
  Safety and tolerability of LY3471851 as assessed through collection of adverse events, serious adverse events, change in vital signs (body temperature, blood pressure, heart rate, rate of breathing and oxygen in blood); electrocardiograms (ECG); laboratory evaluations (hematology, chemistry, liver function and urine analysis).

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Drug Concentration - Time Curve from Zero to the End of Dosing Interval (i.e, 14 days past each dose) (AUC[0-Day 14]) of LY3471851 | Baseline until 14 days after last dose (approximately 43 days after first dose of study drug)
  PK measurement of AUC 0-Day 14
PK: Maximum Observed Drug Concentration (Cmax) of LY3471851 After First and Last Dose | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PK: Measurement of Cmax
PK: Time to Maximum Plasma Concentration (Tmax) of LY3471851 | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PK: Measurement of Tmax
PK: Time to Decrease in Concentration of LY3471851 by Half (T1/2) Due to Elimination | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PK: Measurement of T1/2
Pharmacodynamics (PD): Measurement of Change in Number of Regulatory T Cells (Tregs) and Subsets of Tregs in Blood | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PD: Measurement of Change in Number of Regulatory T Cells (Tregs) and Subsets of Tregs in Blood
PD: Measurement Activity of Tregs | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PD: Measurement Activity of Tregs
PD: Measurement of Change in Number of Subsets of Conventional T Cells (Tcons) in Blood | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PD: Measurement of Change in Number of Subsets of Conventional T Cells
PD: Measurement of Change in Number of Natural Killer Cells (NK Cells) in Blood | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PD: Measurement of Change in Number of Natural Killer Cells (NK Cells) in Blood
PD: Measurement of Cytokines in Blood | Baseline until last study visit (approximately 79 days after first dose of study drug)
  PD: Measurement of Cytokines in Blood
Change in Disease Activity (SLEDAI): Urine; Measurement of Hematuria, Pyuria, Urinary Casts, Creatinine, Protein | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (SLEDAI): Urine; Measurement of Hematuria, Pyuria, Urinary Casts, Creatinine, Protein
Change in Disease Activity (SLEDAI): Blood: Measurement of Anti-dsDNA, Complement, White Blood Cells and Platelets | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (SLEDAI): Blood: Measurement of Anti-dsDNA, Complement, White Blood Cells and Platelets
Change in Disease Activity (Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): Physical Examination | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): Physical Examination
Change in Disease Activity (Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): Urine Analysis | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): Urine Analysis
Change in Disease Activity (Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): Blood Analysis | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Systemic Lupus Erythematosus Disease Activity Index (SLEDAI): Blood Analysis
Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Skin on the Body | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Skin on the Body
Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Mucous Membrane | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Mucous Membrane
Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Scalp | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Scalp
Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Hair Loss | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Cutaneous Lupus Erythematosus Disease Area Severity Index (CLASI): Evaluation of Hair Loss
Change in Disease Activity (Joint score): Evaluation of Tender Joints in the Body | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Joint score): Evaluation of Tender Joints in the Body
Change in Disease Activity (Joint Score): Evaluation of Swollen Joints in the Body | Baseline until last study visit (approximately 79 days after first dose of study drug)
  Change in Disease Activity (Joint Score): Evaluation of Swollen Joints in the Body

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (14):
- United States (14):
  - Investigator Site - Anniston, Anniston, Alabama
  - Investigator Site - La Jolla, La Jolla, California
  - Investigator Site - Clearwater, Clearwater, Florida
  - Investigator Site - Orlando, Orlando, Florida
  - Investigator Site-Tampa, Tampa, Florida
  - Investigator Site - Great Neck, Great Neck, New York
  - Investigator Site- Wilmington, Wilmington, North Carolina
  - Investigator Site - Middleburg Heights, Middleburg Heights, Ohio
  - Investigator Site - Duncansville, Duncansville, Pennsylvania
  - Investigator Site - Jackson, Jackson, Tennessee
  - Investigator Site - Memphis, Memphis, Tennessee
  - Investigator Site - Austin, Austin, Texas
  - Investigator Site - Dallas, Dallas, Texas
  - Investigator Site - Mesquite, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: No